CLINICAL TRIAL: NCT02257203
Title: Evaluation of a Primary Care-Based Intervention to Reduce Consumption of Sugar-sweetened Beverages and 100% Fruit Juice Among Latino Children
Brief Title: Primary Care Beverage Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Academic Pediatric Association (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PC-Based Beverage
Record Dates: First submitted 2014-09-24; First posted 2014-10-06 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Obesity; Dental Caries
Keywords: Dietary sucrose
MeSH Terms: conditions — Obesity; Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar Sweetened Beverage Education (Experimental): Parents will receive an educational module on beverage just after the conclusion of their child's well visit in a private room adjacent to the clinic
  Interventions: Behavioral: Sugar Sweetened Beverage Education
- Reading Education (Active Comparator): Parents will receive an educational module on the importance of reading to children with instruction in interactive reading techniques that are appropriate to the child's age
  Interventions: Behavioral: Reading Education

INTERVENTIONS:
Behavioral: Sugar Sweetened Beverage Education — Parents will receive an educational module on beverage just after the conclusion of their child's well visit in a private room adjacent to the clinic
  Arms: Sugar Sweetened Beverage Education
Behavioral: Reading Education — Parents randomized to control will receive a 25-minute educational module on the importance of reading to children with instruction in interactive reading techniques that are appropriate to the child's age
  Arms: Reading Education

SUMMARY:
This is a pilot randomized clinical trial of a brief educational intervention offered in primary care for Latino parents that promotes healthy beverage consumption by infants and toddlers. The control group will receive an educational intervention that promotes parents reading to children.

DETAILED DESCRIPTION:
To use a randomized controlled trial (RCT) design to test the efficacy of a primary care-based intervention to promote Bright Futures recommendations for consumption of sugar-sweetened beverages and 100% fruit juice among Latino children ages 6 months to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Parents self-identify as Latino
* Parents speak English or Spanish
* Parents have a child between the ages of 6 months and 5 years

Exclusion Criteria:

* Parents who have participated in group educational sessions on nutrition offered through our obesity clinic or who have been newly referred to obesity clinic
* Parents whose child has a chronic condition which affects feeding (such as requiring tube feeds or being on a specialized diet for poor weight gain)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting child's consumption of sugar-sweetened beverages (SSB) | Baseline
  24-hour recall
Number of participants reporting child's consumption of sugar-sweetened beverages (SSB) | 2 weeks
  24-hour recall
Number of participants reporting child's consumption of sugar-sweetened beverages (SSB) | 2 months
  24-hour recall
Number of participants reporting child's consumption of sugar-sweetened beverages (SSB) | 3 months
  24-hour recall
Number of participants reporting child's consumption of 100% fruit juice in excess of guidelines | Baseline
  24-hour recall
Number of participants reporting child's consumption of 100% fruit juice in excess of guidelines | 2 weeks
  24-hour recall
Number of participants reporting child's consumption of 100% fruit juice in excess of guidelines | 2 months
  24-hour recall
Number of participants reporting child's consumption of 100% fruit juice in excess of guidelines | 3 months
  24-hour recall

SECONDARY OUTCOMES:
Servings of SSB and 100% fruit juice in the past 7 days | Baseline
  From the 7-day structured beverage frequency questionnaire we will determine the total servings of SSBs and 100% fruit juice consumed over a 7-day period at each time point
Servings of SSB and 100% fruit juice in the past 7 days | 2 weeks
  From the 7-day structured beverage frequency questionnaire we will determine the total servings of SSBs and 100% fruit juice consumed over a 7-day period at each time point
Servings of SSB and 100% fruit juice in the past 7 days | 2 months
  From the 7-day structured beverage frequency questionnaire we will determine the total servings of SSBs and 100% fruit juice consumed over a 7-day period at each time point
Servings of SSB and 100% fruit juice in the past 7 days | 3 months
  From the 7-day structured beverage frequency questionnaire we will determine the total servings of SSBs and 100% fruit juice consumed over a 7-day period at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Amy L Beck, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Children's Health Center at San Francisco General Hospital, San Francisco, California, United States